CLINICAL TRIAL: NCT03590769
Title: Arterial Imaging of Inflammation and Resolution After Endovascular Surgery
Acronym: AIIRES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-21018
Record Dates: First submitted 2018-05-16; First posted 2018-07-18 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Arterial Disease; Claudication, Intermittent; Claudication; PAD; SFA - Superficial Femoral Artery Stenosis; Iliac Artery Disease; Vascular Calcification
Keywords: Peripheral Arterial Disease; PAD; Claudication, Intermittent; Claudication; SFA Occlusion; Arterial Occlusion; Iliac Artery Occlusion; Vascular Calcification
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Vascular Calcification; Arterial Occlusive Diseases | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Patient undergoing percutaneous angioplasty of SFA or popliteal artery, or stenting of the iliac artery or SFA, will have 18F-FDG-PET scan at the region of interest before intervention, then post-operatively 1 day and 1 week from treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/MR using FDG-18 radiotracer (Experimental): Using FDG-18 radiotracer, subject undergoes PET/MR scan which detects the uptake of the tracer.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All subject will undergo PET/MRI scans pre-operatively, 1 day and 1 week post-operatively using FDG

SUMMARY:
This study evaluates the local inflammatory and resolution response of patients undergoing peripheral vascular intervention like an angioplasty of the superficial femoral artery (SFA) or popliteal artery, or stenting of the iliac artery or SFA, through the use of Positron emission tomography-magnetic resonance imaging (PET/MRI). PET/MRI will be performed prior to intervention, one day and one week after intervention.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) imaging allows for non-invasive visualization of anatomical structures while Positron emission tomography (PET) scans allow for the observation of molecular and cellular activities. Using a PET/MRI in patients with vascular injury post intervention with help evaluate the vascular inflammatory and resolution response in vivo.

Acute vascular injury through endovascular intervention results in recruitment of inflammatory cells such as macrophages to the vessel wall. Macrophages are very metabolically active and consume glucose at a high rate. In PET/MRI, subjects are injected with 18F-Fluorodeoxyglucose (18F-FDG), a radioactively labeled glucose molecule which is consumed by macrophages.

When 18F-FDG is consumed, it is retained within macrophages more avidly than other atherosclerotic lesion elements. Thus, FDG-PET provides a unique and noninvasive approach to quantitatively measure macrophage activity at the intervention site.

This study will provide key pilot data for developing an imaging surrogate endpoint for pro-resolving mediator treatment intervention trials going forward.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 40,
* With resting or exercise ABI <0.9, TBI <0.6
* Have claudication or limb threatening ischemia & planning to undergo a percutaneous angioplasty of SFA or popliteal artery, or stenting of the iliac artery or SFA.

Exclusion Criteria:

* Evidence of active infection
* Hypersensitivity or allergy to contrast agents
* Chronic liver disease, renal disease (GFR< 30) or chronic inflammatory disorders
* Insulin dependent diabetes
* Presence of metal within subject's body, pacemakers, or defibrillators
* BMI < 20 or >35
* Recent other major surgery or illness within 30 days
* Use of immunosuppressive medications or steroids
* History of organ transplantation
* Pregnancy, or plans to become pregnant, or lactating

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Changes found in the quantitative measure of FDG-PET uptake at intervention site prior to and after peripheral vascular injury. | 1 time each week for 3 weeks
  Patient is given 18F-FDG radio tracer. The tracer is quantitatively measured through FDG-PET imaging modality for uptake at the intervention site.

SECONDARY OUTCOMES:
Changes in the correlating the inflammatory and resolution response prior to and after peripheral vascular injury. | 1 time each week for 3 weeks
  Venipuncture of subject and collection of blood allows measures pro-inflammatory markers and targeted metabolipodimics.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Conte, M.D., Principal Investigator — University of California, San Francisco; Miguel H Pampaloni, M.D., PhD., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - UCSF, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong EJ, Chen DC, Westin GG, Singh S, McCoach CE, Bang H, Yeo KK, Anderson D, Amsterdam EA, Laird JR. Adherence to guideline-recommended therapy is associated with decreased major adverse cardiovascular events and major adverse limb events among patients with peripheral arterial disease. J Am Heart Assoc. 2014 Apr 10;3(2):e000697. doi: 10.1161/JAHA.113.000697. PMID 24721799
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Conen D, Rexrode KM, Creager MA, Ridker PM, Pradhan AD. Metabolic syndrome, inflammation, and risk of symptomatic peripheral artery disease in women: a prospective study. Circulation. 2009 Sep 22;120(12):1041-7. doi: 10.1161/CIRCULATIONAHA.109.863092. Epub 2009 Sep 8. PMID 19738135
- [Background] Owens CD, Ridker PM, Belkin M, Hamdan AD, Pomposelli F, Logerfo F, Creager MA, Conte MS. Elevated C-reactive protein levels are associated with postoperative events in patients undergoing lower extremity vein bypass surgery. J Vasc Surg. 2007 Jan;45(1):2-9; discussion 9. doi: 10.1016/j.jvs.2006.08.048. Epub 2006 Nov 21. PMID 17123769
- [Background] Vidula H, Tian L, Liu K, Criqui MH, Ferrucci L, Pearce WH, Greenland P, Green D, Tan J, Garside DB, Guralnik J, Ridker PM, Rifai N, McDermott MM. Biomarkers of inflammation and thrombosis as predictors of near-term mortality in patients with peripheral arterial disease: a cohort study. Ann Intern Med. 2008 Jan 15;148(2):85-93. doi: 10.7326/0003-4819-148-2-200801150-00003. PMID 18195333
- [Background] Carriere I, Dupuy AM, Lacroux A, Cristol JP, Delcourt C; Pathologies Oculaires Liees a l'Age Study Group. Biomarkers of inflammation and malnutrition associated with early death in healthy elderly people. J Am Geriatr Soc. 2008 May;56(5):840-6. doi: 10.1111/j.1532-5415.2008.01677.x. Epub 2008 Apr 9. PMID 18410327
- [Background] Criqui MH, Ho LA, Denenberg JO, Ridker PM, Wassel CL, McDermott MM. Biomarkers in peripheral arterial disease patients and near- and longer-term mortality. J Vasc Surg. 2010 Jul;52(1):85-90. doi: 10.1016/j.jvs.2010.02.004. Epub 2010 May 14. PMID 20471776
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Plasma concentration of C-reactive protein and risk of developing peripheral vascular disease. Circulation. 1998 Feb 10;97(5):425-8. doi: 10.1161/01.cir.97.5.425. PMID 9490235
- [Background] Ridker PM, Stampfer MJ, Rifai N. Novel risk factors for systemic atherosclerosis: a comparison of C-reactive protein, fibrinogen, homocysteine, lipoprotein(a), and standard cholesterol screening as predictors of peripheral arterial disease. JAMA. 2001 May 16;285(19):2481-5. doi: 10.1001/jama.285.19.2481. PMID 11368701
- [Background] Beckman JA, Preis O, Ridker PM, Gerhard-Herman M. Comparison of usefulness of inflammatory markers in patients with versus without peripheral arterial disease in predicting adverse cardiovascular outcomes (myocardial infarction, stroke, and death). Am J Cardiol. 2005 Nov 15;96(10):1374-8. doi: 10.1016/j.amjcard.2005.07.041. Epub 2005 Sep 27. PMID 16275181
- [Background] Tzoulaki I, Murray GD, Lee AJ, Rumley A, Lowe GD, Fowkes FG. C-reactive protein, interleukin-6, and soluble adhesion molecules as predictors of progressive peripheral atherosclerosis in the general population: Edinburgh Artery Study. Circulation. 2005 Aug 16;112(7):976-83. doi: 10.1161/CIRCULATIONAHA.104.513085. Epub 2005 Aug 8. PMID 16087797
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Ho KJ, Spite M, Owens CD, Lancero H, Kroemer AH, Pande R, Creager MA, Serhan CN, Conte MS. Aspirin-triggered lipoxin and resolvin E1 modulate vascular smooth muscle phenotype and correlate with peripheral atherosclerosis. Am J Pathol. 2010 Oct;177(4):2116-23. doi: 10.2353/ajpath.2010.091082. Epub 2010 Aug 13. PMID 20709806
- [Background] Grenon SM, Conte MS, Nosova E, Alley H, Chong K, Harris WS, Vittinghoff E, Owens CD. Association between n-3 polyunsaturated fatty acid content of red blood cells and inflammatory biomarkers in patients with peripheral artery disease. J Vasc Surg. 2013 Nov;58(5):1283-90. doi: 10.1016/j.jvs.2013.05.024. Epub 2013 Jul 2. PMID 23830313
- [Background] Owens CD, Wake N, Conte MS, Gerhard-Herman M, Beckman JA. In vivo human lower extremity saphenous vein bypass grafts manifest flow mediated vasodilation. J Vasc Surg. 2009 Nov;50(5):1063-70. doi: 10.1016/j.jvs.2009.06.022. Epub 2009 Aug 12. PMID 19679424
- [Background] Busti C, Falcinelli E, Momi S, Gresele P. Matrix metalloproteinases and peripheral arterial disease. Intern Emerg Med. 2010 Feb;5(1):13-25. doi: 10.1007/s11739-009-0283-y. Epub 2009 Jul 21. PMID 19626421
- [Background] Brevetti G, Silvestro A, Di Giacomo S, Bucur R, Di Donato A, Schiano V, Scopacasa F. Endothelial dysfunction in peripheral arterial disease is related to increase in plasma markers of inflammation and severity of peripheral circulatory impairment but not to classic risk factors and atherosclerotic burden. J Vasc Surg. 2003 Aug;38(2):374-9. doi: 10.1016/s0741-5214(03)00124-1. PMID 12891123
- [Background] Schillinger M, Exner M, Mlekusch W, Rumpold H, Ahmadi R, Sabeti S, Haumer M, Wagner O, Minar E. Vascular inflammation and percutaneous transluminal angioplasty of the femoropopliteal artery: association with restenosis. Radiology. 2002 Oct;225(1):21-6. doi: 10.1148/radiol.2251011809. PMID 12354979
- [Background] Inoue T, Croce K, Morooka T, Sakuma M, Node K, Simon DI. Vascular inflammation and repair: implications for re-endothelialization, restenosis, and stent thrombosis. JACC Cardiovasc Interv. 2011 Oct;4(10):1057-66. doi: 10.1016/j.jcin.2011.05.025. PMID 22017929
- [Background] Sachs T, Pomposelli F, Hamdan A, Wyers M, Schermerhorn M. Trends in the national outcomes and costs for claudication and limb threatening ischemia: angioplasty vs bypass graft. J Vasc Surg. 2011 Oct;54(4):1021-1031.e1. doi: 10.1016/j.jvs.2011.03.281. Epub 2011 Aug 31. PMID 21880457
- [Background] Mahoney EM, Wang K, Keo HH, Duval S, Smolderen KG, Cohen DJ, Steg G, Bhatt DL, Hirsch AT; Reduction of Atherothrombosis for Continued Health (REACH) Registry Investigators. Vascular hospitalization rates and costs in patients with peripheral artery disease in the United States. Circ Cardiovasc Qual Outcomes. 2010 Nov;3(6):642-51. doi: 10.1161/CIRCOUTCOMES.109.930735. Epub 2010 Oct 12. PMID 20940249
- [Background] Goodney PP, Beck AW, Nagle J, Welch HG, Zwolak RM. National trends in lower extremity bypass surgery, endovascular interventions, and major amputations. J Vasc Surg. 2009 Jul;50(1):54-60. doi: 10.1016/j.jvs.2009.01.035. Epub 2009 May 28. PMID 19481407
- [Background] Havelka GE, Kibbe MR. The vascular adventitia: its role in the arterial injury response. Vasc Endovascular Surg. 2011 Jul;45(5):381-90. doi: 10.1177/1538574411407698. Epub 2011 May 13. PMID 21571779
- [Background] Serhan CN. Pro-resolving lipid mediators are leads for resolution physiology. Nature. 2014 Jun 5;510(7503):92-101. doi: 10.1038/nature13479. PMID 24899309
- [Background] Serhan CN. Resolution phase of inflammation: novel endogenous anti-inflammatory and proresolving lipid mediators and pathways. Annu Rev Immunol. 2007;25:101-37. doi: 10.1146/annurev.immunol.25.022106.141647. PMID 17090225
- [Background] Serhan CN, Yang R, Martinod K, Kasuga K, Pillai PS, Porter TF, Oh SF, Spite M. Maresins: novel macrophage mediators with potent antiinflammatory and proresolving actions. J Exp Med. 2009 Jan 16;206(1):15-23. doi: 10.1084/jem.20081880. Epub 2008 Dec 22. PMID 19103881
- [Background] Oh SF, Pillai PS, Recchiuti A, Yang R, Serhan CN. Pro-resolving actions and stereoselective biosynthesis of 18S E-series resolvins in human leukocytes and murine inflammation. J Clin Invest. 2011 Feb;121(2):569-81. doi: 10.1172/JCI42545. Epub 2011 Jan 4. PMID 21206090
- [Background] Mizwicki MT, Liu G, Fiala M, Magpantay L, Sayre J, Siani A, Mahanian M, Weitzman R, Hayden EY, Rosenthal MJ, Nemere I, Ringman J, Teplow DB. 1alpha,25-dihydroxyvitamin D3 and resolvin D1 retune the balance between amyloid-beta phagocytosis and inflammation in Alzheimer's disease patients. J Alzheimers Dis. 2013;34(1):155-70. doi: 10.3233/JAD-121735. PMID 23186989
- [Background] Chiang N, Fredman G, Backhed F, Oh SF, Vickery T, Schmidt BA, Serhan CN. Infection regulates pro-resolving mediators that lower antibiotic requirements. Nature. 2012 Apr 25;484(7395):524-8. doi: 10.1038/nature11042. PMID 22538616
- [Background] Wang X, Hjorth E, Vedin I, Eriksdotter M, Freund-Levi Y, Wahlund LO, Cederholm T, Palmblad J, Schultzberg M. Effects of n-3 FA supplementation on the release of proresolving lipid mediators by blood mononuclear cells: the OmegAD study. J Lipid Res. 2015 Mar;56(3):674-681. doi: 10.1194/jlr.P055418. Epub 2015 Jan 23. PMID 25616438
- [Background] Recchiuti A, Codagnone M, Pierdomenico AM, Rossi C, Mari VC, Cianci E, Simiele F, Gatta V, Romano M. Immunoresolving actions of oral resolvin D1 include selective regulation of the transcription machinery in resolution-phase mouse macrophages. FASEB J. 2014 Jul;28(7):3090-102. doi: 10.1096/fj.13-248393. Epub 2014 Apr 1. PMID 24692596
- [Background] Hudert CA, Weylandt KH, Lu Y, Wang J, Hong S, Dignass A, Serhan CN, Kang JX. Transgenic mice rich in endogenous omega-3 fatty acids are protected from colitis. Proc Natl Acad Sci U S A. 2006 Jul 25;103(30):11276-81. doi: 10.1073/pnas.0601280103. Epub 2006 Jul 17. PMID 16847262
- [Background] Alie N, Eldib M, Fayad ZA, Mani V. Inflammation, Atherosclerosis, and Coronary Artery Disease: PET/CT for the Evaluation of Atherosclerosis and Inflammation. Clin Med Insights Cardiol. 2015 Jan 7;8(Suppl 3):13-21. doi: 10.4137/CMC.S17063. eCollection 2014. PMID 25674025
- [Background] Rudd JH, Myers KS, Bansilal S, Machac J, Pinto CA, Tong C, Rafique A, Hargeaves R, Farkouh M, Fuster V, Fayad ZA. Atherosclerosis inflammation imaging with 18F-FDG PET: carotid, iliac, and femoral uptake reproducibility, quantification methods, and recommendations. J Nucl Med. 2008 Jun;49(6):871-8. doi: 10.2967/jnumed.107.050294. Epub 2008 May 15. PMID 18483100
- [Background] van der Valk FM, Verweij SL, Zwinderman KA, Strang AC, Kaiser Y, Marquering HA, Nederveen AJ, Stroes ES, Verberne HJ, Rudd JH. Thresholds for Arterial Wall Inflammation Quantified by 18F-FDG PET Imaging: Implications for Vascular Interventional Studies. JACC Cardiovasc Imaging. 2016 Oct;9(10):1198-1207. doi: 10.1016/j.jcmg.2016.04.007. Epub 2016 Sep 14. PMID 27639759
- [Background] Almagor M, Keren A, Banai S. Increased C-reactive protein level after coronary stent implantation in patients with stable coronary artery disease. Am Heart J. 2003 Feb;145(2):248-53. doi: 10.1067/mhj.2003.16. PMID 12595841